CLINICAL TRIAL: NCT04807491
Title: Effects of Kabat Technique and Neuromuscular Re-Education in Patients With Bell's Palsy
Brief Title: Kabat Technique and Neuromuscular Effect in Patients With Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00659 Muhammad Kashif
Record Dates: First submitted 2020-12-21; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; PNF; Kabat therapy; synkinesis
MeSH Terms: conditions — Bell Palsy; Synkinesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kabat Technique's (Active Comparator): Kabat exercises on Upper fulcrum, Intermediate fulcrum and lower fulcrum
  Interventions: Other: Kabat Technique's
- Neuromuscular Re-Education: (Experimental): For initiation, Facilitation, Movement control and movement control
  Interventions: Other: Neuromuscular Re-Education

INTERVENTIONS:
Other: Kabat Technique's — As with all cranial nerves, some specific techniques can also be applied on the facial nerve to enhance responses and improve recovery; the most important are: The rhythmic start: shows and guides the subject into the movements and the scheme; agonist investigation utilizes sequential concentric and eccentric contractions; The inversion of the antagonist: reinforces responses through the induction phenomenon; Repeated contractions: calls for a response with repeated stretching that briefly enables movement; Isometric contractions: for stabilizing and reinforcing the response.
  Conventional therapy exercises
  Arms: Kabat Technique's
Other: Neuromuscular Re-Education — After the baseline assessment, the participant in the control will receive Neuromuscular Re-Education. The duration of session will be 45 minutes.Neuromuscular Re-Education: For initiation (acute phase): Active-assisted exercise,Massage and stretch for affected side.For Facilitation ,Active-assisted exercise.For Movement control:Massage and stretching for facial retraction,Assisted and active exercises on involved side.
  For Relaxation,Thermotherapy,Relaxation exercises,Alternating rhythmic movements.
  Conventional therapy exercises
  Arms: Neuromuscular Re-Education:

SUMMARY:
Bell's palsy is the sudden one-sided peripheral weakness of seventh cranial nerve (Facial nerve), represents 50% to 75% of all etiologies with a rate of 58.2 to 8 new cases per 1 million per year. The objective is to compare the effects of Kabat techniques and Neuromuscular Re-Education on facial disability and synkinesis in patients with bell's palsy. A Randomized Control Trial was conducted on 20 participants, equally allocated in Kabat and PNF training group from February-2020 until December- 2020. Participants were selected according to inclusion and exclusion criteria on purposive sampling technique and randomization was done by sealed envelope method. The assessment was done after taking consent before the first and last session. The tools included Facial disability index, Sunnybrook facial grading system and synkinesis assessment questionnaire. Data were analyzed using SPSS v.20.

DETAILED DESCRIPTION:
Bell's palsy is the sudden one-sided peripheral weakness of seventh cranial nerve (Facial nerve), represents 50% to 75% of all etiologies with the rate of 58.2 to 8 new cases per 1 million per year. It can be either a complete palsy or weakness of facial nerve. This condition may start with pain over half of face especially mastoid region with other symptoms like decreased sensation over half of face, decrease lacrimation, hyperacusis, pain and numbness over half of face. Bell's palsy patients may show signs of absent/decrease facial creases, positive bells phenomenon and forehead folds, associated with other disabilities like contracture in facial muscles and synkinesis due to which patient cannot close his eye.The cause of bell's palsy is unknown therefore it is also called idiopathic facial palsy but recent studies claim that "herpes simplex virus" can be a cause of bell's palsy.Other causes such as tooth extraction, removal of the tumour, local anaesthesia, TMJ surgery, ischemic neuropathy, facial fracture can also be considered. Different studies were carried out on the incidence, risk factors and treatments methods of bell's palsy.The most common risk factors for bell's palsy, reported by a study, is diabetes, and hypertension. A study reported that patients with diabetes are 4 to 5 times more likely to have Bell's palsy.Men and women are equally affected by this disorder.There are different treatment methods for Bells palsy i.e. medical management, physical therapy management, surgical management etc.Although Physical therapy management is not considered to be treatment of choice in treating bell's palsy but there is several clinical studies which claims the benefits of rehabilitation if applied in early stage. Physical therapy managements include different techniques, namely Proprioceptive neuromuscular facilitation, Kabat rehabilitation, Kinisio taping, cryotherapy, massage therapy biofeedback, muscular reeducation.As claimed in a study in 2013, Kabat technique is quite effective in treating the facial disabilities if the therapist is trained. In this study different Kabat techniques namely "rhythmic initiation on those patients who did not perform any movement, repeated stretch was used at the start and also through full ROM in case of muscular weakness, isotonic were used when patients had voluntary movement control, were used on three patients .A study claimed in a case report in 2017 that PNF techniques are very effective in improving functional outcomes in Childs with "bell's palsy".Several studies were done on effects of "Kabat rehabilitation" in "Bell's Palsy". As another conducted a study in 2017.Two groups of Bell's palsy were compared after application of two different treatment protocols. Participants of group A was given Kabat exercises with electrical stimulation and kinesio taping while group B was given electrical stimulation plus home exercises. Study reported that Kabat exercise is quite effective in improving facial asymmetry in bell's palsy.A study was done in 2015 in Islamabad compare the effects of Kabat exercises and Taping in reducing facial synkinesis and disability.The study reported that Kabat exercises are more effective in reducing facial synkinesis and disability.A study was done in 2007, Comparing Neuromuscular reeducation techniques with conventional physical therapy in treating Bell's palsy. This study was done in manipal, India in which he reported that neuromuscular reeducation techniques are more effective in improving facial asymmetry in patients with bell's palsy .The previous studies showed that clinician have worked either with Neuromuscular Re-Education or with kabat in treating Bell's palsy. There is no study done which compare the effects of Neuromuscular Re-Education vs. Kabat in treating Bell's palsy. So the aim of this study is to determine the effect of Kabat and Neuromuscular Re-Education on facial disability and synkinesis and to compare both treatments effects.Kabat Exercises rehabilitation of the facial nerve, 3 fulcrums are found, whose muscles can be stimulated. Upper fulcrum: includes the frontalis, corrugator and orbicularis muscles of the eye.Intermediate fulcrum: Includes the common elevator muscle of the upper lip and wing of nose, the dilator naris and the multiform. Lower fulcrum includes the zygomaticus major, the zygomaticus minor, the risorius, the orbicularis, the triangular of the lower lip, buccinator, chin muscle and square muscle of the chin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of bell's palsy
* Non traumatic onset ( conditions like infectious, hypertensive patients, diabetic patients

Exclusion Criteria:

* • History of significant psychiatric illness

  * Upper motor neuron disease ( stroke, TBI, tumor)
  * Non co-operative patients
  * Post-surgical case

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
SunnyBrook Facial Grading System | 4 weeks
  the tool is used to assess changes from baseline to 4 weeks The Sunnybrook scale is a regional weighted scale based on evaluation of different regions including resting symmetry, symmetry of voluntary movement and severity of Synkinesis to form one single composite score from 0 to 100. It was devised and established at the Sunnybrook Health Sciences Centre in Toronto having an intraclass correlation coefficient (ICC) of 0.890. The Facial Grading System is a tool used for clinical evaluation of Facial Nerve function. It is intended to use on peoples with facial nerve weaknes.

SECONDARY OUTCOMES:
Facial Disability Index | 4 weeks
  the tool is used to assess changes from baseline to 4 weeks The Facial Disability Index (FDI) is a condition-specific scale that is proposed to be used to help clinicians in making decisions about individual patients and to differentiate among individuals with different levels of disability and to evaluate change within a person over time. It have 2 domains, i.e. physical function and social wellbeing. It have total 10 questions, 5/domain. Each item is rated on a 6-point scale, ranging from severe disability to absence of disability. Both subscales are transformed to a score on a 100-point scale, with 100 indicating unimpaired physical or social/well-being function.

OTHER OUTCOMES:
Synkinesis Assessment Questionnair: | 4 weeks
  the tool is used to assess changes from baseline to 4 weeks The Synkinesis Assessment Questionnaire (SAQ) is a valid, reliable, and easily administered instrument for the self-assessment of synkinesis in patients with facial palsy. This instrument was developed and validated in the Facial Nerve Center at the Massachusetts Eye and Ear Infirmary (Boston, USA) in 2007. The questionnaire consists of nine items. Total scores range from 0 (no synkinesis) to 100 (severe synkinesis, all the time). The SAQ is a reliable and valid tool having the Cronbach alpha for the final SAQ was 0.859

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monini S, Iacolucci CM, Di Traglia M, Lazzarino AI, Barbara M. Role of Kabat rehabilitation in facial nerve palsy: a randomised study on severe cases of Bell's palsy. Acta Otorhinolaryngol Ital. 2016 Aug;36(4):282-288. doi: 10.14639/0392-100X-783. PMID 27734980
- [Background] Nicastri M, Mancini P, De Seta D, Bertoli G, Prosperini L, Toni D, Inghilleri M, Filipo R. Efficacy of early physical therapy in severe Bell's palsy: a randomized controlled trial. Neurorehabil Neural Repair. 2013 Jul-Aug;27(6):542-51. doi: 10.1177/1545968313481280. Epub 2013 Apr 2. PMID 23549520
- [Background] Ferreira M, Marques EE, Duarte JA, Santos PC. Physical therapy with drug treatment in Bell palsy: a focused review. Am J Phys Med Rehabil. 2015 Apr;94(4):331-40. doi: 10.1097/PHM.0000000000000255. PMID 25785922
- [Background] Teixeira LJ, Valbuza JS, Prado GF. Physical therapy for Bell's palsy (idiopathic facial paralysis). Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006283. doi: 10.1002/14651858.CD006283.pub3. PMID 22161401
- [Background] Barbara M, Antonini G, Vestri A, Volpini L, Monini S. Role of Kabat physical rehabilitation in Bell's palsy: a randomized trial. Acta Otolaryngol. 2010;130(1):167-72. doi: 10.3109/00016480902882469. PMID 19430987
- [Background] Sardaru D, Pendefunda L. Neuro-proprioceptive facilitation in the re-education of functional problems in facial paralysis. A practical approach. Rev Med Chir Soc Med Nat Iasi. 2013 Jan-Mar;117(1):101-6. PMID 24505900
- [Background] Aranha VP, Samuel AJ, Narkeesh K. Correct the smile of a child by neuromuscular facilitation technique: An interesting case report. Int J Health Sci (Qassim). 2017 Apr-Jun;11(2):83-84. PMID 28539869
- [Background] Manikandan N. Effect of facial neuromuscular re-education on facial symmetry in patients with Bell's palsy: a randomized controlled trial. Clin Rehabil. 2007 Apr;21(4):338-43. doi: 10.1177/0269215507070790. PMID 17613574
- [Background] Mehta RP, WernickRobinson M, Hadlock TA. Validation of the Synkinesis Assessment Questionnaire. Laryngoscope. 2007 May;117(5):923-6. doi: 10.1097/MLG.0b013e3180412460. PMID 17473697
- [Background] Neely JG, Cherian NG, Dickerson CB, Nedzelski JM. Sunnybrook facial grading system: reliability and criteria for grading. Laryngoscope. 2010 May;120(5):1038-45. doi: 10.1002/lary.20868. PMID 20422701
- [Background] Fattah AY, Gurusinghe ADR, Gavilan J, Hadlock TA, Marcus JR, Marres H, Nduka CC, Slattery WH, Snyder-Warwick AK; Sir Charles Bell Society. Facial nerve grading instruments: systematic review of the literature and suggestion for uniformity. Plast Reconstr Surg. 2015 Feb;135(2):569-579. doi: 10.1097/PRS.0000000000000905. PMID 25357164
- [Background] Kleiss IJ, Beurskens CH, Stalmeier PF, Ingels KJ, Marres HA. Synkinesis assessment in facial palsy: validation of the Dutch Synkinesis Assessment Questionnaire. Acta Neurol Belg. 2016 Jun;116(2):171-8. doi: 10.1007/s13760-015-0528-7. Epub 2015 Sep 16. PMID 26377698